CLINICAL TRIAL: NCT02113865
Title: Obtención de un Panel de puntuación ("Score System") Para la predicción de Riesgo Individualizado y la detección Precoz de Carcinoma Hepatocelular (HCC) en Sujetos Coinfectados VIH/VHC
Brief Title: Score System for Prediction Risk and Early Diagnosis of HCC in HIV/HCV Patients
Status: Completed | Type: Observational
Sponsor: Fundacion para la Investigacion Biomedica del Hospital Universitario Ramon y Cajal (Other)
Collaborators: Fundación Mutua Madrileña (Other)
Responsible Party: Sponsor
Other Study IDs: FMM115392013
Record Dates: First submitted 2014-04-07; First posted 2014-04-15 (Estimated); Last update posted 2015-03-09 (Estimated); Status verified 2014-04

CONDITIONS: Acquired Immunodeficiency Syndrome Virus; Hepatitis, Viral, Non-A, Non-B, Parenterally-Transmitted; Hepatocellular Carcinoma
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Hepatitis C; Carcinoma, Hepatocellular

STUDY DESIGN:
Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Serum, plasma, white cells

GROUPS / COHORTS (3):
- Grupo 0: Null or mild fibrosis
- Grupo 1: Cirrhosis
- Grupo 2: HCC diagnosis

SUMMARY:
The aim of this study is to establish a clinical score panel based on clinical, molecular and genetic parameters that allow us to stratify and obtain an early detection of patients with an increased risk of developing hepatocellular carcinoma (HCC).

DETAILED DESCRIPTION:
Transversal study design like a "proof of concept".

Primary objective:

The main objective is try to stablish a descriptive panel (first phase of a score system) based in the conjunction or sum of several clinical and laboratory parameters (molecular and genetic factors). The aim is to detect in a fast, early and successful way those patients that presents a high risk to develop an hepatocellular carcinoma (HCC) in the future in a specific population: HIV and HCV coinfected patients. The establishment of this panel will allow clinicians set up a correct treatment decreasing the probability of liver cirrhosis and HCC.

ELIGIBILITY:
Inclusion Criteria:

* Human immunodeficiency virus chronic infection
* Hepatitis C virus chronic infection
* No other liver viral coinfections

Exclusion Criteria:

* Alcohol consume
* Immunosuppressor or immunoactive treatment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV/HCV coinfected patients from Infectious Diseases Department
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2013-10; Primary Completion 2014-10 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Sera inflammatory markers | 1 day (Routine visit to normal following in Infectious Disease Department)
  Inflammatory markers will be measure used a Enzyme-linked Immunosorbent Assay

SECONDARY OUTCOMES:
Sera apoptotic markers | 1 day (Routine visit in disease following at Infectious Disease Department)
  Apoptotic markers will be evaluated through a Enzyme-linked Immunosorbent Assay

OTHER OUTCOMES:
Evaluation of genetic polymorphisms distribution between study groups of relevant genes probably implicated in the disease | 1 day (Routine visit in normal following at Infectious Disease Department)
  Genetic polymorphisms will be evaluated using Real-Time polymerase chain reaction technique

CONTACTS AND LOCATIONS:
Overall Officials: Beatriz S Sastre, PhD, Principal Investigator — Fundación para la Investigación Biomédica del Hospital Ramón y Cajal
Locations (1):
- Hospital Ramón y Cajal, Madrid, Spain